CLINICAL TRIAL: NCT05774340
Title: A Randomized, Double-Blind, Placebo-Controlled Phase Ⅱ Clinical Study to Evaluate the Efficacy and Safety of CM326 in Subjects With Moderate to Severe Asthma
Brief Title: A Study of CM326 in Subjects With Moderate to Severe Asthma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM326-001
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-03

CONDITIONS: Moderate to Severe Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CM326 Low Dose (Experimental): CM326 220 mg/2 mL, subcutaneous at low dose
  Interventions: Drug: CM326
- CM326 High Dose (Experimental): CM326 220mg/2mL, subcutaneous at high dose
  Interventions: Drug: CM326
- Placebo (Placebo Comparator): Placebo 2mL, subcutaneous
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CM326 — CM326 injection
  Arms: CM326 High Dose; CM326 Low Dose
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a multi-center, randomized, double-blind, placebo-controlled Phase Ⅱ clinical study to evaluate the efficacy, safety, PK characteristics, PD effects and immunogenicity of CM326 in subjects with moderate to severe asthma.

The study consists of three periods, including an up to 4-week screening period, a 52-week treatment period, and a 12-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the study and voluntarily sign the informed consent form.
2. Age ≥18 and ≤75 years old, male or female, weight ≥40 kg.
3. The subject has been diagnosed with asthma for at least 1 year.
4. Pre-bronchodilator FEV1 measured ≤80% of the normal predicted value.
5. A positive bronchodilation test within 24 months before informed consent or at screening.
6. The subject has received medium-to-high dose ICS combined with at least one control drug, such as LABA, LAMA, LTRA, theophylline, for at least 3 months before signing the informed consent, and maintained stable treatment regimen and dosage for at least 1 month before signing the informed consent.
7. Asthma Control Questionnaire-5 (ACQ-5) score ≥1.5.
8. Subjects must have experienced at least one severe asthma exacerbation event within 12 months before informed consent, and have not experienced a severe asthma exacerbation event within 1 month before informed consent.
9. Subjects (including partners) have no plans to have children and voluntarily use highly effective contraception from the time of signing the informed consent form until 3 months after the last dose.

Exclusion Criteria:

1. Received biological agents with the same therapeutic purpose within 6 months before signing the informed consent.
2. Prior autoimmune disease or inflammatory treatment with biologic agents/systemic immunosuppressive agents within 8 weeks or 5 half-lives (whichever is longer) prior to informed consent.
3. Received immune globulin or blood products within 30 days before informed consent.
4. Subjects treated with systemic corticosteroids other than for the treatment of asthma from 8 weeks before signing the informed consent to the date of randomization.
5. Received live or attenuated vaccine within 3 months before informed consent signing or planned to receive live or attenuated vaccine during the study period.
6. Initiation of desensitization therapy within 3 months before informed consent.
7. Underwent bronchial thermoplasty within 12 months before informed consent.
8. Current smokers or former smokers who quit smoking less than 6 months or former smokers who quit smoking more than 6 months with a smoking history of more than 10 pack-years.
9. Chronic obstructive pulmonary disease (COPD) or other lung disease that may impair lung function, as judged by the investigator.
10. Active infection or acute infection requiring systemic anti-infective therapy from 4 weeks before enrollment to the time of randomization.
11. Previous history of known or suspected immunosuppression, including a history of invasive opportunistic infection, even if the infection has resolved; or the presence of unusual frequent, recurrent, or prolonged infections.
12. History of malignancy.
13. The presence of any severe and/or uncontrolled medical condition that in the judgment of the investigator may affect the evaluation of the drug, including but not limited to: severe neurological disease, history of severe mental disorder, major cardiovascular disease, diabetes mellitus poorly controlled by intensive treatment, QTcF interval prolongation, or persistent arrhythmia.
14. Major surgery within 8 weeks prior to informed consent or planned surgery requiring general anesthesia or hospitalization for > 1 day during the study period.
15. Fertile women with positive pregnancy test results during screening; pregnant or lactating women.
16. Positive screening serologic test for HIV or treponema pallidum.
17. Chronic hepatitis B virus or hepatitis C virus infection.
18. Subjects with abnormal liver and kidney function, such as aspartate aminotransferase or alanine aminotransferase>2× ULN, or serum creatinine>1.5× ULN.
19. Have systemic diseases other than asthma that result in an elevated peripheral blood eosinophil count or other diseases such as helminth parasitic infections for which standard treatment is not received or does not respond.
20. Allergy or intolerance to components of CM326 injection or placebo or history of severe drug allergy or anaphylactic shock.
21. Have been enrolled in a clinical trial of any drug or medical device within 3 months before signing informed consent, or are within the follow-up period of a clinical study or the five half-lives of the trial drug (whichever is longer) before signing informed consent.
22. Subjects who have used heavy alcohol within 3 months before screening.
23. History of drug abuse within 5 years before signing informed consent.
24. The investigator considers that there are any conditions that may prevent the subject from completing the study or present a significant risk to the subject or other factors that may reduce the likelihood of enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of subjects experiencing severe asthma exacerbations | 24 weeks
  Annualized rate of subjects experiencing severe asthma exacerbations during the 24-week randomized treatment period.

SECONDARY OUTCOMES:
Annualized rate of subjects experiencing the event of loss of asthma control (LOAC) | 24 weeks
  Annualized rate of subjects experiencing the event of loss of asthma control (LOAC) during the 24-week randomized treatment period.
Change from baseline in pre-bronchodilator forced expiratory volume in 1 second (FEV1) | 64 weeks
  Change from baseline in pre-bronchodilator FEV1 at each evaluation time point.
Rate of change from baseline in pre-bronchodilator FEV1 | 64 weeks
  Rate of change from baseline in pre-bronchodilator FEV1 at each evaluation time point.
Time to the first onset of the severe asthma exacerbation event | 52 weeks
  Time from baseline to the first onset of the severe asthma exacerbation event.
Time to the onset of the first event of LOAC | 52 weeks
  Time from baseline to the onset of the first event of LOAC.
Change from baseline in FEV1 percentage of predicted value (FEV1% Pred) | 64 weeks
  Change from baseline in FEV1% Pred at each evaluation time
Change from baseline in Peak diurnal and nocturnal expiratory flow (PEF) | 64 weeks
  Change from baseline in PEF at each evaluation time
Change from baseline in Forced vital capacity (FVC) | 64 weeks
  Change from baseline in FVC at each evaluation time
Change from baseline in Forced Expiratory Flow (FEF) 25-75% | 64 weeks
  Change from baseline in 25-75%FEF at each evaluation time
Change from baseline in FEV1 after the use of bronchodilator | 64 weeks
  Change from baseline in FEV1 after the use of bronchodilator at each evaluation time
Change from baseline in the Asthma Control Questionnaire-5 (ACQ-5) score at each evaluation time point | 64 weeks
  Change from baseline in the ACQ-5 score at each evaluation time point
Change from baseline in asthma symptom score at each evaluation time point | 64 weeks
  Change from baseline in asthma symptom score at each evaluation time point
Change from baseline in the Standardized Asthma Quality of Life Questionnaire (AQLQ(S)) score at each evaluation time point | 64 weeks
  Change from baseline in the AQLQ(S) score at each evaluation time point
Change from baseline in the number of inhalations of SABA | 64 weeks
  Change from baseline in the number of inhalations of SABA at each evaluation time
Incidence of Adverse events (AEs) | 64 weeks
  Incidence of AEs, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.
Pharmacokinetic profile of CM326 | 64 weeks
  Maximum Plasma Concentration（Cmax）of CM326
Immunogenicity | 64 weeks
  Incidence of anti-drug antibodies (ADAs) and neutralizing antibodies (Nabs) (if applicable).

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided